CLINICAL TRIAL: NCT06847373
Title: Efecto De La Suplementación De Vitamina D En La Resistencia a La Insulina En Escolares Y Adolescentes Con Obesidad
Brief Title: Efficacy and Safety of Vitamin D Supplementation in Pediatric Patients with Obesity
Acronym: VD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-2022-3603-018
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Vitamin D; Insulin Resistance; Obesity, Childhood
Keywords: vitamin D; insulin resistence; obesity; leptin; adiponectin; pediatric
MeSH Terms: conditions — Insulin Resistance; Pediatric Obesity; Obesity | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Intervention Model Description: randomized double-blind clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cholecalciferol 4000UI (Vitamin D) (Experimental): 4000 IU daily orally during six months.
  Interventions: Dietary Supplement: Cholecalciferol
- Cholecalciferol 1000U (Vitamin D) (Sham Comparator): 1000 IU daily orally during six months. .
  Interventions: Dietary Supplement: Cholecalciferol

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — cholecalciferol 4000 IU daily orally
  Other Names: Vitamin D

SUMMARY:
Introduction: Vitamin D deficiency is commonly observed in patients with obesity, primarily due to sequestration by adipose tissue. Recent research highlights the importance of this deficiency, showing a correlation between low vitamin D levels and mechanisms contributing to insulin resistance.

Objectives: This study aims to compare the effects of supplementing with 4,000 IU of vitamin D versus 1,000 IU over six months on insulin resistance and the leptin/adiponectin ratio in school-aged children and adolescents with obesity.

Materials and Methods: A controlled clinical trial will be conducted involving 40 children with obesity aged 10 to 18 years (BMI >95th percentile). Participating children and their parents will undergo measurements such as weight, height, BMI, body fat, and Tanner stage. All participants will receive dietary and physical activity recommendations based on WHO guidelines. After initial assessments, participants will be randomly assigned to receive either 4,000 IU or 1,000 IU of vitamin D. They will be monitored monthly for capsule intake and adverse effects, with follow-up measurements of anthropometry, leptin, adiponectin, insulin & lipid profile.

Statistical Analysis: Baseline characteristics will be compared using t-Student or U-Mann Whitney tests, depending on variable distribution. The intervention's impact will be assessed by calculating deltas for body fat and biochemical measurements, with significance tested using paired t-tests or Wilcoxon tests. Covariance analysis (ANCOVA) will be used to adjust for confounding variables.

DETAILED DESCRIPTION:
Materials and Methods The study will compare the effect of 4000 IU vitamin D supplementation over six months on adipokines (leptin/adiponectin ratio) and insulin resistance (HOMA index) in school-aged children and adolescents with obesity, against a similar group receiving 1000 IU of vitamin D. The study will be conducted at the Hospital Infantil de México Federico Gómez and UMAE Hospital de Pediatría, Centro Médico Nacional Siglo XXI. This controlled clinical trial features an experimental, randomized, double-blind design. The study population includes schoolchildren with obesity attending the Adolescent Clinic at Hospital Infantil de México and outpatient services at UMAE Hospital de Pediatría.

Sampling and Selection Criteria A non-probabilistic sampling will select children identified with obesity. Selection criteria include both male and female patients aged 10 to 18 with obesity as per BMI (>95th percentile according to WHO age and sex tables), who agree to participate, and reside in Mexico City. Exclusion criteria exclude patients with comorbidities unrelated to obesity, genetic syndromes, those currently receiving vitamin supplements or pharmacological treatments for obesity, and those with pre-existing insulin resistance requiring pharmacological treatment.

Treatment Arms Group A will receive 4000 IU of vitamin D daily for six months. Group B, the control group, will receive 1000 IU daily. Randomization is managed using a software tool, with treatment assignments sealed in opaque envelopes and administered according to randomized allocation.

Sample Size and Statistical Analysis Sample size calculations for unpaired group comparisons anticipate 20 participants per group, adjusting for a 20% dropout rate, based on differences in the leptin/adiponectin ratio and HOMA index. Statistical analyses will be performed on both an intention-to-treat and per-protocol basis. Descriptive analysis will evaluate quantitative variables' distribution using the Kolmogorov-Smirnov test to determine appropriate statistical tests. Comparative analyses will utilize t-tests or U-Mann Whitney tests for quantitative variables, and chi-squared or Fisher's exact tests for categorical data. Mixed-effects regression models will assess changes in dependent variables over time. Analyses will be conducted using Stata version 14.0, with a confidence level of ≤0.05.

Procedures and Follow-Up Prior to the intervention, patients will undergo comprehensive assessments including anthropometry and blood tests. Dietary and physical activity plans will be provided, tailored to each patient's caloric needs and physical capabilities. Monthly follow-ups will ensure adherence to the supplementation regimen and monitor any adverse effects. The final assessment will repeat all initial evaluations to assess changes after six months of treatment.

Blinding and Data Integrity The study ensures blinding for medical staff, patients, families, and data collectors. The treatment capsules for both groups will be identical in appearance to maintain blinding integrity throughout the trial.

Study Conclusion The study concludes with a final collection of anthropometric and blood sample data after six months, which will be analyzed to determine the effectiveness of vitamin D supplementation on improving insulin resistance and adipokine levels among children and adolescents with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants.
* Participants aged between 10 and 18 years.
* Obesity as defined by a Body Mass Index (BMI) in the >95th percentile according to the World Health Organization's age and sex-specific tables.
* Willingness to participate in the study.
* Residency in Mexico City.

Exclusion Criteria:

* Patients with comorbidities not attributable to obesity, such as chronic kidney disease, heart failure, liver cirrhosis, etc.
* Patients with Prader-Willi syndrome, Albright's hereditary osteodystrophy, Borjesson-Forssman-Lehmann syndrome.
* Patients currently taking vitamin supplements.
* Patients undergoing pharmacological treatment for obesity.
* Patients who already present insulin resistance and, although they have not previously received medication, are currently indicated for pharmacological treatment with metformin.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in 25 hydroxi vitamin D at 6 Months. | From enrollment to the end of treatment at 6 months
  A peripheral blood sample will be collected. Patients are required to fast for 12 hours prior to presenting for blood sample collection, scheduled between 7:00 and 8:00 AM. Blood will be drawn via venipuncture and subsequently centrifuged at 3000 revolutions per minute for five minutes to separate the serum. The serum will be aliquoted and stored at -20 degrees Celsius until further analysis. The levels of 25-hydroxy Vitamin D will be quantified using an ELISA method, employing the 6913 25(OH) Vitamin D ELISA Kit (96 Tests - Abcam) in conjunction with the Varioskan™ LUX multimode microplate reader.
  At the end of the six-month study, a second blood sample will be collected to assess vitamin D levels at that time.
  Vitamin D Concentration Standards:
  Normal: Greater than 30 ng/mL Insufficiency: 20-30 ng/mL Deficiency: Less than 20 ng/mL
Change from Baseline in leptin at 6 Months. | From enrollment to the end of treatment at 6 months
  A sample of peripheral blood will be collected to measure serum levels of leptin. Patients are required to fast for 12 hours and should arrive for the sample collection between 7:00 and 8:00 AM. The blood will be drawn through venipuncture. After collection, the sample will be centrifuged at 3000 revolutions per minute for five minutes. The serum will then be aliquoted for subsequent analyses. These serum samples will be stored at -20 degrees Celsius until they are analyzed. Leptin will be measured using the ELISA technique with the commercial kit from Merck Millipore, Milliplex Map Human Adipokine Magnetic Bead Panel Endocrine Multiplex Assay.
  At the end of the six-month study, a second blood sample will be collected to assess leptin levels at that time.
Change from Baseline in adiponectin at 6 Months. | From enrollment to the end of treatment at 6 months
  A sample of peripheral blood will be collected to measure serum levels of adiponectin. Patients are required to fast for 12 hours and should arrive for the sample collection between 7:00 and 8:00 AM. The blood will be drawn through venipuncture. After collection, the sample will be centrifuged at 3000 revolutions per minute for five minutes. The serum will then be aliquoted for subsequent analyses. These serum samples will be stored at -20 degrees Celsius until they are analyzed. Adiponectin will be measured using the ELISA technique with the commercial kit from Merck Millipore, Milliplex Map Human Adipokine Magnetic Bead Panel Endocrine Multiplex Assay.
  At the end of the six-month study, a second blood sample will be collected to assess adiponectin levels at that time.
Change from Baseline in insulin at 6 Months. | From enrollment to the end of treatment at 6 months
  Insulin is an anabolic hormone secreted by the pancreas that plays a role in regulating blood glucose level. A sample of peripheral blood will be collected to measure serum levels of insulin . Patients are required to fast for 12 hours and should arrive for the sample collection between 7:00 and 8:00 AM. The blood will be drawn through venipuncture. After collection, the sample will be centrifuged at 3000 revolutions per minute for five minutes. The serum will then be aliquoted for subsequent analyses. These serum samples will be stored at -20 degrees Celsius until they are analyzed. Insulin levels will be determined through the chemiluminescence technique using the Varioskan™ LUX multimode microplate reader. At the end of the six-month study, a second blood sample will be collected to assess insulin levels at that time.
Change from Baseline in HOMA-IR at 6 Months. | From enrollment to the end of treatment at 6 months
  The HOMA-IR index is utilized to evaluate the relationship between glucose and insulin, assessing insulin resistance. It is calculated using the formula: HOMA = (Glucose * Insulin) / 405. At the end of the six-month study, At the end of the six-month study, the HOMA-IR index will be calculated again.
Change from Baseline in triglycerides at 6 Months. | From enrollment to the end of treatment at 6 months
  Triglycerides, a class of lipids, consist of one glycerol molecule bonded to three fatty acids. To determine triglyceride levels, a sample of peripheral blood will be collected from patients who must fast for 12 hours and arrive for sampling between 7:00 and 8:00 AM. The blood will be drawn through venipuncture, then centrifuged at 3000 revolutions per minute for five minutes, and the serum will be separated into aliquots for analysis. These samples will be stored at -20 degrees Celsius until tested. Triglyceride concentrations will be measured using a colorimetric method on the Varioskan™ LUX multimode microplate reader, an automated clinical chemistry analyzer. Triglyceride levels below 100 mg/dL in children under 10 years and below 130 mg/dL in individuals over 10 years are considered abnormal. At the end of the six-month study, a second blood sample will be collected to assess triglyceride levels at that time.
Change from Baseline in HDL cholesterol at 6 Months. | From enrollment to the end of treatment at 6 months
  High-density lipoprotein (HDL) cholesterol consists of smaller and denser lipoproteins, composed of a high proportion of proteins, and acts as a protective factor against cardiovascular disease. To determine HDL cholesterol levels, a peripheral blood sample will be collected from patients who are required to fast for 12 hours and arrive for sampling between 7:00 and 8:00 AM. Blood will be drawn through venipuncture, then centrifuged at 3000 revolutions per minute for five minutes. The serum will be separated into aliquots for subsequent analysis. These samples will be stored at -20 degrees Celsius until they are tested. HDL cholesterol levels will be measured using a colorimetric method on the Varioskan™ LUX multimode microplate reader, an automated clinical chemistry analyzer. Normal values are considered to >40 mg/dL. At the conclusion of the six-month study, a second blood sample will be collected to reassess the HDL cholesterol levels.
Change from Baseline in LDL cholesterol at 6 Months. | From enrollment to the end of treatment at 6 months
  To determine Low-density lipoprotein (LDL) cholesterol, a peripheral blood sample will be collected from patients required to fast for 12 hours and arrive for sampling between 7:00 and 8:00 AM. Blood will be drawn via venipuncture and then centrifuged at 3000 revolutions per minute for five minutes. The serum will be separated into aliquots for subsequent analysis. These samples will be stored at -20 degrees Celsius until they are tested. LDL cholesterol levels will be measured using a colorimetric method on the Varioskan™ LUX multimode microplate reader, an automated clinical chemistry analyzer. Levels considered abnormal are >130 mg/dL.
  At the end of the six-month study period, a second blood sample will be collected to reassess the LDL cholesterol levels.
Change from Baseline in total cholesterol at 6 Months. | From enrollment to the end of treatment at 6 months
  Total cholesterol is an essential molecule vital for life, performing crucial structural and metabolic functions in the human body. To measure total cholesterol levels, a peripheral blood sample will be collected from patients who must fast for 12 hours and arrive for sampling between 7:00 and 8:00 AM. Blood will be drawn through venipuncture, then centrifuged at 3000 revolutions per minute for five minutes. The serum will be separated into aliquots for further analysis. These samples will be stored at -20 degrees Celsius until they are tested. Total cholesterol levels will be determined using a colorimetric method with the Varioskan™ LUX multimode microplate reader, an automated clinical chemistry analyzer. Normal total cholesterol levels are considered to be less than 200 mg/dL.
  At the conclusion of the six-month study, a second blood sample will be collected to reassess total cholesterol levels.
Change from Baseline in glucose at 6 Months. | From enrollment to the end of treatment at 6 months
  Glucose is a vital molecule that provides energy to the body. To measure glucose levels, a peripheral blood sample will be collected from patients who must fast for 12 hours and arrive for sampling between 7:00 and 8:00 AM. Blood will be drawn through venipuncture, then centrifuged at 3000 revolutions per minute for five minutes. The serum will be separated into aliquots for further analysis. These samples will be stored at -20 degrees Celsius until they are tested. Glucose levels will be determined using a colorimetric method with the Varioskan™ LUX multimode microplate reader, an automated clinical chemistry analyzer.
  At the conclusion of the six-month study, a second blood sample will be collected to reassess glucose levels.
Change from Baseline in The Body Mass Index at 6 Months. | From enrollment to the end of treatment at 6 months
  The Body Mass Index (BMI): A measure of the relationship between an individual's weight and height. It will be determined using the formula: weight (kg) / height^2 (m²). At the end of the six-month study, the BMI will be recalculated.
Change in the Z-score of the Body Mass Index at 6 Months. | From enrollment to the end of treatment at 6 months
  The Z-score of the Body Mass Index (BMI) is a statistical measurement that expresses the number of standard deviations a person's BMI is from the mean or average BMI of a population. This score is particularly useful in pediatric populations to assess how a child's body mass compares to that of their peers, considering age and gender.
  The calculation is based on national or global reference data that standardizes BMI according to age and sex. This standardized score helps to accurately identify and categorize underweight, healthy weight, overweight, and obesity in children and adolescents. At the start of the study, the BMI Z-score will be calculated to establish baseline levels for each participant. At the end of the six-month study period, the BMI Z-score will be recalculated to determine any changes.
Change in the leptin/adiponectin ratio at 6 months | From enrollment to the end of treatment at 6 months
  The leptin/adiponectin ratio represents the ratio of serum leptin to adiponectin levels. It will be determined through laboratory analysis after a 12-hour fasting period. Leptin and adiponectin will be measured using the ELISA technique with the commercial kit from Merck Millipore, Milliplex Map Human Adipokine Magnetic Bead Panel Endocrine Multiplex Assay.Following the 6-month study period, a second blood sample will be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil de Mexico Federico Gomez, México, Mexico